CLINICAL TRIAL: NCT00134693
Title: A Randomised, Placebo-controlled, Parallel Group Single Dose Study of SB681323 in Patients With Active RA to Investigate the CRP Dose Response Relationship
Brief Title: A Single Dose Of Compound SB-681323 Compared To Prednisolone On A Protein That Is an Indicator For Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA1104046
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: SB-681323 rheumatoid arthritis CRP biomarkers
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisolone; dilmapimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Prednisolone
Drug: SB-681323
  Other Names: Prednisolone

SUMMARY:
This study is designed to compare a range of doses of SB-681323 with prednisolone, which has known effects on rheumatoid arthritis patients. By comparing the two drugs and their effects on blood proteins that indicate for rheumatoid arthritis, we hope to ascertain information on the most effective dose of SB-681323 to use in future.

ELIGIBILITY:
Inclusion criteria:

* Must have a diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology.
* Must have 3 or more swollen or 3 or more tender/painful joints at screening.
* Must be on stable weekly methotrexate (2.5mg - 25mg) for at least eight weeks prior to screening.

Exclusion criteria:

* Must not be morbidly obese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-06-21 (Actual); Primary Completion 2006-08-03 (Actual); Study Completion 2006-08-03 (Actual)

PRIMARY OUTCOMES:
Analysis for C-Reactive protein (CRP) levels 72 hours post-dose following SB-681323 | Day 3 (at 72 hour)
  CRP levels were compared between SB-681323 and placebo 72 hours post-dose. The ratio of the dose response relationship of placebo and 7.5mg, 15mg and 25mg of SB-681323 has been presented.

SECONDARY OUTCOMES:
Analysis of CRP levels 24 and 48 hours post-dose following SB-681323 | Day 1 (at 24 hour) and Day 2 (at 48 hour)
  CRP levels were compared between SB-681323 and placebo 24 and 48 hours post-dose. The ratio of the dose response relationship of placebo and 7.5mg, 15mg and 25mg of SB-681323 has been presented.
Analysis of Interleukin (IL)-6 levels up to 72 hours post-dose following SB-681323 | Upto Day 3 (at 1, 3, 24 and 72 hour)
  A blood sample of approximately 5 milliliter (mL) was taken for measurement of serum markers. IL-6 measurements were performed at 1 hour, 3, hours, 24 hours and 72 hours post-dose. The ratio of the dose response relationship of placebo and 7.5mg, 15mg and 25mg of SB-681323 has been presented.
Number of participants with adverse events (AE) and serious adverse events (SAE) | Upto Day 3 (72 hours)
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury. There were no SAEs reported in this study.
Change from Baseline in vital sign systolic blood pressure (SBP) and diastolic blood pressure (DBP) | Baseline (at pre-dose Day 0) and Day 3 (at 90 minutes, 3 hour, 24 and 72 hour)
  Supine vital signs SBP and DBP were recorded whilst the participant was in a supine position (participant lying flat with maximum one pillow) having rested in that position for at least 10 minutes before each reading. Measurements were performed at 90 minutes, 3 hours, 24 hours and 72 hours post-dose. Baseline was defined as assessment performed pre-dose at Day 0. Change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization values at the time of assessment.
Change from Baseline in vital sign heart rate | Baseline (at pre-dose Day 0) and Day 3 (at 90 minutes, 3 hour, 24 and 72 hour)
  Supine vital signs (heart rate) was recorded whilst the participant was in a supine position (participant lying flat with maximum one pillow) having rested in that position for at least 10 minutes before each reading. Measurements were performed at 90 minutes, 3 hours, 24 hours and 72 hours post-dose. Baseline was defined as assessment performed pre-dose at Day 0. Change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization values at the time of assessment.
Number of participants with abnormal electrocardiogram (ECG) findings | Day 1 (pre-dose, 1 hour and 3 hour)
  Full 12-lead ECGs were recorded using an ECG machine that automatically calculated the pulse rate and measured PR, RR, QRS, QT, QTc(b) intervals (Bazett's correction was applied to QTc measurements). Measurements were carried out at pre-dose, 1 hour and 3 hours on Day 1. ECG findings were characterized as abnormal-not clinically significant (A-NCS) and abnormal-clinically significant (A-CS). Data has been presented for A-NCS findings on Day 1.
Number of participants with clinical chemistry data outside the clinical concern range | Upto Day 3 (pre-dose, 24, 48 and 72 hours
  Clinical chemistry parameters included albumin, alkaline phosphatase, alanine amino transferase, indirect bilirubin, calcium, chloride, creatinine, gamma glutamyl transferase, glucose, potassium, lactate dehydrogenase, triglycerides. Measurements were carried out at pre-dose, 24 hours, 48 hours and 72 hours. Data for number of participants with values outside clinical concern range defined as high and low have been presented.
Number of participants with hematology data outside the clinical concern | Upto Day 3 (pre-dose, 24 and 72 hours)
  Hematology parameters included eosinophils, hemoglobin, hematocrit, lymphocytes, mean corpuscle hemoglobin, mean corpuscle volume, platelet count, reticulocytes, white blood cell count (WBC). Measurements were carried out at pre-dose, 24 hours and 72 hours. Data for number of participants with values outside clinical concern range defined as high and low have been presented.
Number of participants with abnormal urinalysis dipstick results | Upto Day 3 (pre-dose, 24 and 72 hours)
  Approximately 10-20 mL mid-stream urine was collected into a sterile container and was screened by dipstick for: occult blood, proteins, ketones, glucose, red blood cells (RBC) and WBC. Sediment microscopy was performed only if any of the Multi-stick tests were abnormal. In such cases, microscopy was performed for: WBC, RBC, hyaline casts, granular casts, cellular casts. Data for number of participants with abnormal urinalysis results for positive parameters as assessed by dipstick and microscopic analysis have been presented.
Whole blood messenger RNA (mRNA) levels of tumor necrosis factor alpha [TNF-α], IL-8, IL-1β and Cyclo-oxygenase-2 [COX-2] (and other genes implicated in the pathogenesis of RA or genes involved in the mode of action of the compounds administered) | Pre-dose, 45 minutes, 90 minutes and 3 hours on Day 1
  Blood samples were taken for extraction of whole blood mRNA (2 x 2.5mL PAXgene tubes). The samples were taken at the time-points pre-dose, 45 minutes, 90 minutes and 3 hours. Messenger RNA levels for various markers was measured. These markers included Prednisolone markers: DDIT4, DUSP1, FKBP5, GILZ, IL1R2, TXNIP, ZNF145 and p38 markers: COX2, IFI30, IL1b, IL6, IL8, TNF. An aliquot of mRNA was stored for later analysis of other genes associated with the pathogenesis of RA and in the mode of action of the compounds administered.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- Australia (7):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Douglas, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Daw Park, South Australia
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Shenton Park, Western Australia
- France (2):
  - GSK Investigational Site, Amiens, Picardie
  - GSK Investigational Site, Montpellier
- Germany (5):
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- United Kingdom (6):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Wigan, Lancashire
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Newcastle, Northumberland
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Sheffield